CLINICAL TRIAL: NCT02895789
Title: Evaluation of Oxidative Capacity and Exercise Tolerance in Ambulatory Patients With Spinal Muscular Atrophy (SMA)
Brief Title: Oxidative Capacity and Exercise Tolerance in Ambulatory SMA
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Jacqueline Montes, Assistant Professor of Rehabilitation and Regenerative Medicine , Rehab & Regenerative Med PT, Columbia University
Other Study IDs: AAAQ9447; 1K01HD084690-01A1 (NIH)
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Spinal Muscular Atrophy Type 3; Mitochondrial Myopathy
Keywords: spinal muscular atrophy; oxidative capacity; exercise tolerance; mitochondrial myopathy; SMA; six minute walk test; neuromuscular disease; ambulation; exercise; mitochondria; cycle ergometry; near infrared spectroscopy
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Mitochondrial Myopathies; Muscular Atrophy, Spinal; Neuromuscular Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- spinal muscular atrophy: ambulatory children and adults ages between 8 and 55 years old by the time of enrollment with laboratory documentation of homozygous deletion of SMN1 exon 7
- mitochondrial myopathy: ambulatory children and adults ages between 8 and 55 years old by the time of enrollment with genetic confirmation or evidence from muscle biopsy confirming the diagnosis
- control: The healthy control group will be age and gender-matched to the SMA and mitochondrial myopathy groups as best as possible.

SUMMARY:
This proposal will focus on (1) estimating oxidative capacity of specific muscle groups during exercise using near infrared spectroscopy and (2) describing body composition to better understand exercise capacity and mitochondrial function in ambulatory spinal muscular atrophy (SMA) patients and disease controls. It is a 6-month observational study including 14 ambulatory SMA patients, 14 ambulatory patients with mitochondrial myopathy, and 14 healthy controls.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is a progressive, recessively-inherited neuromuscular disease characterized by weakness and muscle atrophy due to the loss of spinal cord motor neurons. The results from this study would provide preliminary data, using non-invasive methods, on oxidative capacity in ambulatory SMA patients and disease controls to aid in the design of exercise intervention studies. Furthermore, this information would link previous laboratory and preclinical findings of mitochondrial depletion in SMA to the clinical condition and provide important information for future studies designed to improve oxidative capacity and fitness in SMA patients.

ELIGIBILITY:
Inclusion Criteria:

1. One of the following categories:

   * Genetic confirmation of SMA with laboratory documentation of homozygous deletion of SMN1 exon 7;
   * Genetic confirmation of mitochondrial myopathy or evidence from muscle biopsy confirming the diagnosis; or
   * Healthy individuals.
2. Able to walk independently at least 25 meters, and able to tread a stationary cycle ergometer.

Exclusion Criteria:

1. Unable to walk 25 meters independently.
2. Use of investigational medications intended for the treatment of SMA within 30 days prior to study entry.
3. The presence of any contraindication to exercise according the ACSM criteria.

Patients with and without Spinraza treatment are eligible.

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study sample will include 14 ambulatory SMA patients, 14 ambulatory mitochondrial myopathy patients, and 14 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Change in NIRS derived index of muscle oxygen extraction | baseline, 6 months
  Near Infrared Spectroscopy (NIRS) is a simple, non-invasive method to measure oxygen in muscle and other tissues in vivo.

SECONDARY OUTCOMES:
Change in Peak oxygen uptake (V02 max) | baseline, 6 months
  Participants will undergo an exercise stress test performed by a clinical exercise physiologist using an electronically-braked recumbent cycle ergometer to determine peak oxygen uptake (VO2 max).
Change in Distance walked during the Six Minute Walk Test (6MWT) | baseline, 6 months
  6MWT is an objective evaluation of functional exercise capacity, measures the maximum distance a person can walk in six minutes over a 25-meter linear course.
Change in Lean body mass assessed with Dual Energy X-ray Absorptiometry (DEXA) | baseline, 6 months
  Dual-Energy X-ray Absorptiometry (DEXA) is a method of estimating bone and lean body mass by comparing the absorption of two distinct energy level beams at 46.8 keV and 80 keV, which are effective at differentiating soft tissue and bone. A standard DEXA scan will be performed in supine.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Montes, PT, EdD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided